CLINICAL TRIAL: NCT03459586
Title: The Purpose of This Study is to Determine if the 9zest App for Parkinson's Disease (PD) is Feasible, Safe, and Efficacious When Used Independently by Individuals With Parkinson's Disease
Brief Title: A Mobile Application for Telerehabilitation in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: 9zest. Inc. (Industry)
Collaborators: University of Nevada, Las Vegas (Other); Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9zest parkinson study
Record Dates: First submitted 2018-02-24; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to determine if the 9zest app for Parkinson's disease is feasible, safe, and efficacious when used independently by individuals with Parkinson's disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 9zest app facilitated exercise (Experimental): App to facilitate exercises for 3 times a week for 12 weeks. The app includes physical therapist-designed exercises that are modified using an algorithm to the participants physical capabilities and PD status. Exercises include strengthening, balance, range of motion, and endurance type exercise.
  Interventions: Other: 9zest app facilitated exercise

INTERVENTIONS:
Other: 9zest app facilitated exercise — The purpose of this study is to determine if the 9zest app for Parkinson's disease is feasible, safe, and efficacious when used independently by individuals with Parkinson's disease

SUMMARY:
The purpose of this study is to determine if the 9zest app for Parkinson's disease is feasible, safe, and efficacious when used independently by individuals with Parkinson's disease.

DETAILED DESCRIPTION:
The investigators will evaluate the 9zest app using a non-randomized, single-group design wherein participants who have downloaded the 9zest app will be informed via a message in the app about the trial and invited to participate. If the participant answers yes to the invitation the participant will be consented through a questionnaire in the app. In the consent form for participation, prospective participants will learn the eligibility criteria. If the participant completes the informed consent process, the participant will then be required to answer specific inclusion and exclusion criteria questions to ensure qualification for the study. A phone number that goes directly to a member of the research team will be provided if the prospective participant has any questions during the informed consent process.

Outcome measurements. After completing the consent process and prior to participation in the 12-week trial, participants will answer several questions about specific symptoms to complete their registration and profile. The participant will then be asked to perform a couple of pretest outcome measures via the app. Participants will also be tested at the 4 week, 8 week, and 12 week marks.

Exercise intervention. The 12-week app guided exercise intervention is a personalized exercise regimen. Participants will use the smartphone/tablet app for the study period of 12 weeks. While the app has been developed to deliver physical therapy in a variety of movement disorders including multiple system atrophy, progressive supranuclear palsy, and dementia with Lewy bodies, users will choose the PD track for the purposes of the study, which is the population of interest. The participants will create a PD profile with a series of questions to assess the current level of functioning. A proprietary algorithm (9zest Smart™) developed by physical therapists and information technologists chooses the appropriate workout regimen for the person's level of function. The customized regimen is intended to be safe and effective for the participant. The 9zest App Family has over 1,000 original therapy videos in its library, which encompasses Physical Therapy, Fitness, Yoga, Meditation, and Speech Therapy. 9zest Smart™, the app's intelligent engine determines the right set and levels of exercises for a user based on the Smart Assessment responses. At preset intervals (generally after 2 weeks), the app will again assess the user's functional capacity and needs. Again, the 9zest Smart algorithm will adjust the type, duration, and intensity of the regimen to maximize performance. All of the exercises and dosing features are consistent with contemporary and evidence-based physical therapy practice. Additionally, the exercises have all been deemed to be safe by physical therapists for each particular level of function. The exercise program is imbedded in the app. A demonstration of the exercise is shown in audiovisual format and then the participant follows along with the exercise in real time.

Participants in the trial will be asked to participate in the 12-week exercise program with the goal of participating 3 times per week with each session lasting 60 minutes. After the trail is over, the investigators will sort and analyze the data based on compliance (eg, high engagers, moderate engagers, low engagers).

ELIGIBILITY:
Inclusion Criteria:

* English speaking men and women between 40 and 75 years old
* Neurologist-diagnosed PD
* A caregiver who is willing to assist the participant
* Willingness to participate is a 12 week study
* Be able to stand unassisted for 10 minutes
* Stable on PD medication and deep brain stimulation for 3 months prior to trial

Exclusion Criteria:

* Failure on a cognition screen
* Co-morbidities that would preclude exercise participation or increase participant risk: severe osteoarthritis/pain, stroke, severe respiratory problems, traumatic brain injury, neuromuscular disease, atrial fibrillation, poorly controlled cardiovascular disease, limb amputation, osteoporosis)
* Vision or hearing impairment that would interfere with app use
* Fall that required physician evaluation (ED, urgent care, hospitalization) with the past year
* Use of an assistive device (or person) for walking, standing, balance.
* Currently use of a structured exercise regimen defined as participation in a regular exercise program consisting of more than 60 minutes per week in total

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and falls during exercise using the 9 zest app | 12 week measurement point
  At the end of the trial, the investigators will analyze the incidence of exercise-related adverse events and falls that occurred while exercising using the 9 zest app over the course of the study. These adverse events will be self-reported using a questionnaire and will be analyzed using frequencies, means, and measures of variability.
Self-report questionnaire on the feasibility and usability of exercising using the 9 zest app | 12 week measurement point
  A 5 point Likert style, self-report questionnaire with 6 items taken from the Intrinsic Motivation Inventory will be used to examine ease of use, design, user friendliness of exercising while using the 9zest app. Each of the 6 items will be reported separately. Scores range from 1 to 5 for each item.

SECONDARY OUTCOMES:
The change in the number of times a participant can go from sitting to standing in 30 seconds | Change in score from pretest to 3 posttests (4 week, 8 week, and 12 week measurement points)
  The 30 second Sit-To-Stand test will be used to determine a signal of efficacy for functional lower extremity strength.
The change in the amount of time a person can go from a sitting position to walking 3 meters, turning around and going back to sitting. | Change in score from pretest to 3 posttests (4 week, 8 week, and 12 week measurement points)
  The Timed Up and Go Test will be used for a signal of efficacy regarding dynamic gait performance.
The change in score on a self-report questionnaire of quality of life regarding mobility | Change in score from pretest to 3 posttests (4 week, 8 week, and 12 week measurement points)
  The Parkinson's Disease Questionnaire-39 mobility subscale has 10 disease-specific mobility-related questions and will be used to determine a signal of efficacy related to disease-specific mobility. Each of the 10 items has a 5 item Likert response with scores ranging from 0 to 4. The scores of all 10 items will be added up and divided by the total possible points (40 points); thus, this outcome measurement will be reported as a percent of the total possible points with a lower score being suggestive of higher mobility-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Merrill Landers, DPT, PhD, Principal Investigator — UNLV, Las Vegas
Locations (1):
- Merrill Landers, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Landers MR, Ellis TD. A Mobile App Specifically Designed to Facilitate Exercise in Parkinson Disease: Single-Cohort Pilot Study on Feasibility, Safety, and Signal of Efficacy. JMIR Mhealth Uhealth. 2020 Oct 5;8(10):e18985. doi: 10.2196/18985. PMID 33016887